CLINICAL TRIAL: NCT05890339
Title: Laparoscopic Proximal Gastrectomy With Double-flap Technique Versus Laparoscopic Total Gastrectomy With Roux-en-Y Reconstruction for Proximal Early Gastric Cancer: a Multi-center Randomized Controlled Trial
Brief Title: Laparoscopic Proximal Gastrectomy With Double-flap Technique Versus Laparoscopic Total Gastrectomy With Roux-en-Y Reconstruction for Proximal Early Gastric Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: First Hospital of China Medical University (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Liaoning Cancer Hospital & Institute (Other); Sichuan Provincial People's Hospital (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Qilu Hospital of Shandong University (Other); First Affiliated Hospital of Kunming Medical University (Other); First Affiliated Hospital of Guangxi Medical University (Other); Zunyi Medical College (Other); Sichuan Cancer Hospital and Research Institute (Other); Gansu Provincial Hospital (Other); Shandong Provincial Hospital (Other Government); The First Affiliated Hospital of Zhengzhou University (Other); Qinghai Province Cancer Hospital (Unknown); LanZhou University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2022-276-02
Record Dates: First submitted 2023-05-03; First posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2022-09

CONDITIONS: Stomach Neoplasms
Keywords: laparoscopy; minimally invasive surgical procedures; stomach neoplasm; Gastrectomy; Reflux Esophagitis
MeSH Terms: conditions — Stomach Neoplasms; Esophagitis, Peptic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic Proximal Gastrectomy With Double-flap Technique (Experimental)
  Interventions: Procedure: Laparoscopic Proximal Gastrectomy With Double-flap Technique
- Laparoscopic Total Gastrectomy With Roux-en-Y Reconstruction (Active Comparator)
  Interventions: Procedure: Laparoscopic Total Gastrectomy With Roux-en-Y Reconstruction

INTERVENTIONS:
Procedure: Laparoscopic Proximal Gastrectomy With Double-flap Technique — Patients in this group receive laparoscopic proximal gastrectomy with D1+/D2 lymph node dissection(D1+ for stage IA：Nos.1, 2, 3a, 4 sa, 4 sb, 7, 8a, 9, 11p；D2 for stage IB: Nos.1, 2, 3a, 4 sa, 4 sb, 7, 8a, 9, 11p and 11d). The double-flap technique is used for the esophagogastric reconstruction.
  Arms: Laparoscopic Proximal Gastrectomy With Double-flap Technique
Procedure: Laparoscopic Total Gastrectomy With Roux-en-Y Reconstruction — Patients in this group receive laparoscopic total gastrectomy with D1+/D2 lymph node dissection(D1+ for stage IA：Nos.1, 2, 3, 4, 5, 6, 7, 8a, 9, 11p；D2 for stage IB: Nos.1, 2, 3, 4, 5, 6, 7, 8a, 9, 11p and 11d, 12a). The Roux-en-Y esophagojejunostomy method is used for the esophagojejunal reconstruction.
  Arms: Laparoscopic Total Gastrectomy With Roux-en-Y Reconstruction

SUMMARY:
Proximal early gastric cancer can choose radical total gastrectomy or proximal gastrectomy. But if use simple esophagogastric anastomosis for proximal gastrectomy, the incidence of postoperative reflux esophagitis is up to 62%, which seriously affects the quality of life, and the short-term outcome is poorer than the total gastrectomy. If the incidence of postoperative reflux esophagitis can be reduced, proximal gastrectomy would be the treatment choice for proximal early gastric cancer, which may more improve both quality of life and nutritional status than total gastrectomy.

Double-flap technique is a new surgical procedure for the reconstruction between esophagus and remnant stomach, which was started to be applied to digestive tract reconstruction in patients with proximal early gastric cancer in 2016. It can reduce the occurrence of reflux oesophagitis. At present, the studies for double-flap technique in China and other countries are mostly retrospective studies, and there are short of large-scale prospective studies and evidence of evidence-based medicine.

The applicant has initiated a phase II, single center, single arm study and the results suggested that the laparoscopic proximal gastrectomy with double-flap reconstruction technique was safe and effective for treating proximal early gastric cancer. To further validate the short and long-term outcomes of this procedure, a multicentre, open label, prospective, superiority and randomised controlled clinical trial was set up to compare laparoscopic proximal gastrectomy with double-flap technique with laparoscopic total gastrectomy with Roux-en-Y reconstruction for proximal early gastric cancer. It include 216 patients with proximal early gastric cancer. The primary outcome is the proportion of patients who develop reflux esophagitis within 12 months after surgery. The short and long-term oncological outcomes are also explored. This trial can provide high-grade evidence of evidence-based medicine for double-flap technique's clinical applications .

ELIGIBILITY:
Inclusion Criteria:

1. 20 years ≤ age ≤ 80 years
2. The primary gastric lesions were located in the proximal third of the stomach
3. histologically proven gastric adenocarcinoma (by preoperative gastrofiberscopy)
4. clinical stage IA (T1N0M0) or IB (T1N1M0 / T2N0M0) according to the 8th edition of the American Joint Committee on Cancer(AJCC) staging system(Clinical stage was determined based on the finding of endoscopic ultrasonography and/or thoraco-abdominal contrast-enhanced computed tomography)
5. scheduled for laparoscopic proximal gastrectomy with D1+/D2 lymphadenectomy or laparoscopic total gastrectomy with D1+/D2 lymphadenectomy , and possible for R0 surgery by this procedures (Lymphadenectomy is performed on the basis of the criteria of the Japanese Gastric Cancer Treatment Guidelines 2021 (6th edition).).
6. The preoperative American Society of Anesthesiologists (ASA) physical status was I-III; The patient's cardiopulmonary function can tolerate laparoscopic surgery.
7. The patients have signed the informed consent form.

Exclusion Criteria:

1. history of upper abdominal surgery (except laparoscopic cholecystectomy);
2. the tumor invades the esophagus 3cm above gastro-esophageal junction (Z-line)
3. with other malignant diseases or have suffered from other malignant diseases within 5 years
4. require simultaneous surgery due to complicated with other diseases
5. women are pregnant or in lactation period
6. Suffering from serious mental illness
7. history of continuous systemic corticosteroid or immunosuppressive drug treatment within 1 month

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2023-06-10 (Estimated); Primary Completion 2029-12-10 (Estimated); Study Completion 2033-05-10 (Estimated)

PRIMARY OUTCOMES:
The Proportion of Patients With Reflux Esophagitis Within 12 Months Postoperatively | 12 months postoperatively
  During follow-up endoscopy 1 year after surgery, reflux esophagitis are graded according to the Los Angeles (LA) classification.

SECONDARY OUTCOMES:
Quality of Life after Surgery | Follow-up evaluations are performed 3, 6 and 12 months postoperatively
  Quality of life(QoL) is evaluated using the European Organization for Research and Treatment of Cancer (EORTC) 30-item core QoL (QLQ-C30 ver.3.0). Higher scores mean a worse outcome.
Gastrointestinal Symptoms after Surgery | Follow-up evaluations are performed 3, 6 and 12 months postoperatively
  gastrointestinal symptoms are assessed by Gastrointestinal Quality of Life Index (GIQLI) questionnaires. Higher scores mean a better outcome.
Changes in hemoglobin levels at Follow-up | Follow-up evaluations are performed 3, 6 and 12 months postoperatively.
  blood hemoglobin(g/L) levels
Changes in Vitamin B12 levels at Follow-up | Follow-up evaluations are performed 3, 6 and 12 months postoperatively.
  blood Vitamin B12（μg/ml) levels
Changes in total protein levels at Follow-up | Follow-up evaluations are performed 3, 6 and 12 months postoperatively.
  blood total protein(g/L) levels
Changes in serum albumin levels at Follow-up | Follow-up evaluations are performed 3, 6 and 12 months postoperatively.
  blood serum albumin(g/L) levels
Changes in prealbumin levels at Follow-up | Follow-up evaluations are performed 3, 6 and 12 months postoperatively.
  blood prealbumin(g/L) levels
Late Postoperative Morbidity | Follow-up evaluations are performed 3, 6 and 12 months postoperatively.
  adhesive ileus, anastomosis stenosis, malnutrition, dumping syndrome. All postoperative complications are classified according to the Clavien-Dindo(CD) classification standard.
Early Postoperative Morbidity | From surgery to discharge, up to 30 days
  operation wound with seroma, hematoma, infection, dehiscence, or evisceration, anastomotic leakage, anastomotic bleeding, abdominal bleeding, abdominal abscess, intestinal obstruction morbidity, gastrointestinal bleeding, gastroparesis, postoperative pancreatitis, pancreatic fistula, chylous leakage, lung morbidity, cerebrovascular morbidity, cardiovascular morbidity, deep vein thrombosis, cholecystitis, liver dysfunction, kidney dysfunction. All postoperative complications are classified according to the Clavien-Dindo(CD) classification standard.
Short-term Clinical Outcome After Surgery | From surgery to discharge, up to 30 days
  time to pass gas(hours)
Short-term Clinical Outcome After Surgery | From surgery to discharge, up to 30 days
  time to oral intake(hours)
Short-term Clinical Outcome After Surgery | From surgery to discharge, up to 30 days
  time to indwell gastric tube(hours)
Short-term Clinical Outcome After Surgery | From surgery to discharge, up to 30 days
  length of postoperative hospitalisation(days)
Surgical Characteristics | 24 hours postoperatively
  operative time(minutes)
Surgical Characteristics | 24 hours postoperatively
  time for reconstruction the digestive tract(minutes) during surgery
Surgical Characteristics | 24 hours postoperatively
  blood loss(ml) during surgery
3-year disease-free survival rate | 3 years
  3-year disease-free survival rate
3-year overall survival rate | 3 years
  3-year overall survival rate
3-year recurrence pattern | 3 years
  3-year recurrence pattern
5-year disease-free survival rate | 5 years
  5-year disease-free survival rate
5-year overall survival rate | 5 years
  5-year overall survival rate
5-year recurrence pattern | 5 years
  5-year recurrence pattern
body mass index postoperatively | Follow-up evaluations are performed 3, 6 and 12 months postoperatively.
  body mass index(kg/m^2)
Quality of Life postoperatively | Follow-up evaluations are performed 3, 6 and 12 months postoperatively
  Quality of life(QoL) is evaluated using the European Organization for Research and Treatment of Cancer (EORTC) gastric cancer module (QLQ-STO22) questionnaire. Higher scores mean a worse outcome.
Postoperative pain assessment | Day 1 postoperatively
  We measured the pain score using visual analog scale(VAS) at 24 hours after the surgery is completed. Higher scores mean a worse outcome.
Pathological Characteristics | 1 week postoperatively
  lymph nodes dissection extent for each patient in the surgery
Pathological Characteristics | 1 week postoperatively
  number of dissected lymph nodes for each patient in the surgery
Pathological Characteristics | 1 week postoperatively
  R0 resection rate. R0 resection represents complete resection of the tumor, meaning there is no residual tumor.
Proportion of participants die after surgery | From surgery to discharge, up to 30 days
  mortality rate
Proportion of participants need to rehospitalized after surgery | From surgery to discharge, up to 30 days
  rehospitalization rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zhou S, Xie Y, Zhu Y, Tan J, Yang B, Zhong L, Zhong G, Han F. Comparing the antireflux effect of laparoscopic proximal gastrectomy with double-flap technique reconstruction versus laparoscopic total gastrectomy with Roux-en-Y reconstruction for proximal early gastric cancer: study protocol for a multicentre, prospective, open-label, randomised controlled trial. BMJ Open. 2024 Jul 4;14(7):e079940. doi: 10.1136/bmjopen-2023-079940. PMID 38964794